CLINICAL TRIAL: NCT02386527
Title: Consortium of Early Arthritis Cohorts USA - A Prospective Cohort Study of Adults With New Consent Inflammatory Arthritis Symptoms to Understand Predictors of Optimal Outcomes
Brief Title: Consortium of Early Arthritis Cohorts USA
Acronym: CATCH-US
Status: Terminated | Type: Observational
Why Stopped: This study has been terminated by PI and BRANY IRB on 4/18/24.
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Northwestern University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Vivian Bykerk, MD, Hospital for Special Surgery, New York
Other Study IDs: 2014-229
Record Dates: First submitted 2015-02-26; First posted 2015-03-12 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Maximum of 7 tubes of blood will be collected
Oversight: Data Monitoring Committee: No

SUMMARY:
Rheumatoid arthritis (RA) is the most common form of inflammatory arthritis. In the US, it is estimated that as many as 3 million adults may suffer from the disease. Fortunately in the last few years, a shift in strategy toward the earlier institution of disease modifying drugs and the availability of new classes of medications have greatly improved the outcomes that can be expected by most patients.

The goal of treatment now aims toward achieving the lowest possible level of arthritis disease activity and even remission, if possible as early on as possible. Research has shown that this translates into minimized joint damage and enhanced physical function and quality of life for the RA patient. This also requires that a diagnosis of RA be made as early on as possible, and herein lies the challenge, i.e. identifying the RA patient early on in the course of their disease.

DETAILED DESCRIPTION:
This is a study of usual care, a prospective cohort of all eligible and consenting patients referred to the Inflammatory Arthritis Center of Excellence and the Division of Rheumatology, Department of Medicine at HSS as well as 3 consortium sites across the U.S.

In order to study the effectiveness of recommended treatments in usual practice in different patients for short-term and long-term outcomes, and to determine factors that may predict how a patient's disease might progress over time, investigators will need to analyze and describe the strategies used to manage these patients and will need to understand:

i. The frequency of single time-point and sustained (two or more time points) remission or low disease activity over time ii. Factors that influence remission iii. Which patients can achieve persistent sustained remission, and iv. Who can undergo drug withdrawal and still sustain remission of low disease activity v. Factors associated with treatment optimization or barriers to achieving this

ELIGIBILITY:
Inclusion Criteria:

* Patient was 18 years of age or over at time of referral
* Joint symptoms for < 12 months
* 2+ swollen joints OR 1 swollen joint with one of the following: Rheumatoid Factor > 20 IU, (+) anti-CCP antibody, morning stiffness > 45 minutes, responded to NSAIDs, (+) MTP squeeze test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Most patients will have been referred by their primary care providers (PCP) for an expedited assessment and all will have met inclusion criteria. If the patient is appropriate for inclusion into the cohort, the study will be explained to the patient by the rheumatologist or designate. If he/she is interested, the information sheet and consent form will be reviewed with the study nurse or coordinator and consent will be obtained. As this is a study of usual care, study data is the information collected during regular clinic visits. Therefore, the patient will be consenting to have the data from their regular assessments entered into the study database. A schedule of regular visits has been identified in advance in keeping with best clinical practice and management of ERA.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Rapidity and sustainability of SDAI remission as achieved over a one year period | 3 months, 6 months, 9 months and 12 months of follow-up

SECONDARY OUTCOMES:
The proportion of patients achieving DAS28 remission and CDAI remission twice | 3 months, 6 months, 9 months and 12 months of follow-up
Rapid radiographic progression, as measured by a van der Heijde Sharp Score change of 5 point or more | 2 months and 24 months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States